CLINICAL TRIAL: NCT03246217
Title: Efficacy of Therapeutic Instrumental Music Performance With Sensory-Enhanced Motor Imagery in Improving Therapeutic Outcomes for Individuals With Chronic Post-Stroke Hemiparesis
Brief Title: Therapeutic Instrumental Music Performance With Sensory-Enhanced Motor Imagery in Chronic Post-Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Catherine Haire, PhD Candidate, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #34521
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic Instrumental Music Performance (Experimental): Therapeutic Instrumental Music Performance is a Neurologic Music Therapy technique in which selection of instruments, spatial configurations and sequences for playing are designed to facilitate retraining of movement patterns used in everyday life. Participants will receive nine individual forty-five minute sessions of Therapeutic Instrumental Music Performance, three sessions per week.
  Interventions: Behavioral: Therapeutic Instrumental Music Performance
- Therapeutic Performance with Sensory-Enhanced Motor Imagery (Experimental): Participants will receive nine individual sessions, three times per week: thirty minutes of Therapeutic Instrumental Music Performance, followed by fifteen minutes of sensory-enhanced motor imagery. During sensory-enhanced motor imagery, participants will listen to a metronome set to their preferred pace for previously practised movements while engaging in motor imagery.
  Interventions: Behavioral: Therapeutic Instrumental Music Performance; Behavioral: Therapeutic Performance with Sensory-Enhanced Motor Imagery
- Therapeutic Performance with Motor Imagery (Experimental): Participants will receive nine individual sessions, three times per week: thirty minutes of Therapeutic Instrumental Music Performance, followed by fifteen minutes of motor imagery. Motor imagery will involve mental practice of previous movement exercises.
  Interventions: Behavioral: Therapeutic Instrumental Music Performance; Behavioral: Therapeutic Performance with Motor Imagery

INTERVENTIONS:
Behavioral: Therapeutic Instrumental Music Performance — Participants will play a variety of instruments (acoustic and electronic) to facilitate retraining of everyday functional movements.
Behavioral: Therapeutic Performance with Sensory-Enhanced Motor Imagery — Participants will listen to a metronome set to their preferred pace for previously practised movements while engaging in motor imagery.
  Arms: Therapeutic Performance with Sensory-Enhanced Motor Imagery
Behavioral: Therapeutic Performance with Motor Imagery — Participants will engage in motor imagery of previously practised movements.
  Arms: Therapeutic Performance with Motor Imagery

SUMMARY:
Research has shown that music engages the brain bilaterally throughout cortical and subcortical regions, accessing extended sensorimotor, cognitive and affective networks. This research explores the hypothesis that use of these shared neural networks allows neurologic music therapy interventions targeting upper extremity motor control to promote plasticity and functional improvements in persons recovering from a cerebrovascular accident. The potential therapeutic benefits of these interventions on attentional processes and affective responding will also be examined.

DETAILED DESCRIPTION:
More individuals are surviving and living with the effects of stroke, a trend that is expected to continue. Upper extremity limitations present a common, persistent challenge for stroke survivors, impacting quality of life. In addition, links have been found between physical impairment and depression, and depression and stroke-induced cognitive impairment. Music has been shown to exert multimodal effects on individuals and may be used as a mediating stimulus to promote therapeutic change. Furthermore, motor imagery may enhance the effectiveness of upper extremity interventions by engaging the same brain areas that are active in physical movement. The purpose of this study is to investigate the effects of therapeutic instrumental music performance and sensory-enhanced motor imagery on upper limb movement, affect and cognition following a stroke. Participants will be assessed at two baselines, and randomly assigned to one of three intervention groups: therapeutic instrumental music performance, therapeutic instrumental music performance and sensory-enhanced motor imagery, or therapeutic instrumental music performance and motor imagery without sensory enhancement.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis following a unilateral stroke (hemorrhagic or ischemic), sustained more than 6 months prior, with at least minimal volitional movement of the affected limb
* permission from a physician to participate in an upper extremity rehabilitation program, including confirmation that the following disorders are not present: rheumatoid arthritis, upper extremity fracture, apraxia, neuropathy, somatosensory impairment
* adequate language comprehension and neurocognitive function to understand and follow simple instructions

Exclusion Criteria:

* currently enrolled in an upper extremity rehabilitation program or another upper extremity study
* comorbid neurological disorder (e.g. multiple sclerosis, Parkinson's disease)
* evidence of perceptual or cognitive impairment; e.g., unilateral spatial neglect, significant hearing impairment, Montreal Cognitive Assessment score of 25 or less
* presence of aphasia
* injections for spasticity within three months of participation

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Wolf Motor Function Test | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Measures upper extremity motor ability through timed and functional tasks.
Changes from baseline in Fugl-Meyer Assessment Upper Extremity | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Performance based measure assessing motor capacity.

SECONDARY OUTCOMES:
Motor Activity Log | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Individuals rate quality and amount of movement during daily functional tasks.
Trunk Impairment Scale | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Assessment of upper trunk impairment using the upper trunk items of the Trunk Impairment Scale
Multiple Affect Adjective Check List-Revised | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Measure of affective state
General Self-Efficacy Scale | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Assessment of perceived self-efficacy
Digit Span | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Assesses working memory and attention
Trail Making Test Part B | Baseline 1, Baseline 2 (1 week later), Post intervention of 4 weeks
  Assesses mental flexibility and processing speed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thaut, PhD, Principal Investigator — University of Toronto
Locations (1):
- Faculty of Music, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loria T, de Grosbois J, Haire C, Vuong V, Schaffert N, Tremblay L, Thaut MH. Music-based intervention drives paretic limb acceleration into intentional movement frequencies in chronic stroke rehabilitation. Front Rehabil Sci. 2022 Oct 3;3:989810. doi: 10.3389/fresc.2022.989810. eCollection 2022. PMID 36262914